CLINICAL TRIAL: NCT03913611
Title: A Randomised Controlled Trial of Accelerated Rehabilitation Versus Standard Rehabilitation After Double-row Rotator Cuff Repair. Does Rehabilitation Regimen Affect Clinical Outcomes?
Brief Title: Shoulder Surgery Traditional vs Accelerated Rehabilitation Trial
Acronym: S-START
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSTART
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Tear or Rupture, Not Specified as Traumatic
Keywords: Shoulder arthroscopy; Rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to two groups, with balanced numbers entering each group.
Who Masked: Outcomes Assessor
Masking Description: The therapist assessing patients' range of movement and the radiologist assessing integrity of the repair will be blinded to the arm of the trial that the patient entered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Rehabilitation (Other): In this arm, patients will undergo the standard rehabilitation protocol, with sling use for 6 weeks.
  Interventions: Other: Traditional rehabilitation protocol
- Accelerated Rehabilitation (Experimental): In this arm, patients will undergo the accelerated rehabilitation protocol, with no sling use outside the immediate postoperative period.
  Interventions: Other: Accelerated rehabilitation protocol

INTERVENTIONS:
Other: Accelerated rehabilitation protocol — Patients in this group will undergo an accelerated rehabilitation protocol, without movement restrictions. Movement restriction will instead be governed by patient comfort.
  Arms: Accelerated Rehabilitation
Other: Traditional rehabilitation protocol — Patients in this group will undergo a traditional rehabilitation protocol, with movement restrictions and sling use for 6 weeks following surgery.
  Arms: Traditional Rehabilitation

SUMMARY:
This is a randomised controlled trial involving patients who have a double-row arthroscopic rotator cuff repair.

Null hypothesis: There is no difference in outcome between standard rehabilitation and accelerated rehabilitation after arthroscopic rotator cuff repair.

Following surgery, they will be randomised to one of two groups:

1. Standard rehabilitation, with enforced sling use for 6 weeks and a structured exercise programme.
2. Accelerated rehabilitation with no requirement to use a sling and a structured exercise programme.

The primary outcome measure will be the Oxford Shoulder Score at 6 months. We will also collect data on postoperative pain, range of shoulder movement and other subjective outcome measures. All patients will have MRI scans at 6 months postoperatively to assess the integrity of the repair, allowing comparison of failure rates between groups.

DETAILED DESCRIPTION:
This is a randomised controlled trial involving patients who have a double-row arthroscopic rotator cuff repair. We wish to compare clinical and radiological outcomes for patients undergoing standard rehabilitation protocols versus accelerated rehabilitation.

A double-row repair will be used in this study as it has been shown in laboratory testing to be stronger and withstand significantly more cyclical loads before failure.

Patients who have failed conservative treatment for their rotator cuff tears will be offered inclusion in the study. Baseline scores and measurements will be taken prior to surgery. After a successful surgical repair has been confirmed, patients will be randomised to one of two rehabilitation programmes. One programme will mandate use of a sling for 6 weeks, and another will not require use of a sling after the immediate postoperative period.

All patients will be followed up for one year, at intervals of 6 weeks, 3 months, 6 months and 12 months, using subjective outcome measures, objective measures of movement and an MRI scan to assess the integrity of the repair at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 40 with a degenerate full-thickness posterosuperior rotator cuff tear undergoing arthroscopic rotator cuff repair (+/- concomitant procedures such as biceps tenotomy and subacromial decompression).

Exclusion Criteria:

* Other musculoskeletal disease affecting same limb
* Massive rotator cuff tear
* Subscapularis tear
* Incomplete cuff repair
* Repair under tension
* Non-English speaker
* Inability to follow postoperative instructions / restrictions

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 3 months
  A validated patient-reported outcome measure of shoulder function. This score ranges from 0-48, with higher scores representing a better outcome.

SECONDARY OUTCOMES:
Oxford Shoulder Score | 6 weeks, 3 months, 6 months, 12 months postoperatively.
  A validated patient-reported outcome measure of shoulder function. This score ranges from 0-48, with higher scores representing a better outcome.
Shoulder Pain and Disability Index | 6 weeks, 3 months, 6 months, 12 months postoperatively.
  A validated patient-reported outcome measure of shoulder function. This score is composed to two subscales. One is for pain and the other subscale is for disability. Both subscales range from 0 to 100, with lower scores representing a better outcome. The scores are averaged to provide a global score.
EQ5D | 6 weeks, 3 months, 6 months, 12 months postoperatively.
  A validated patient-reported outcome measure of general health. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This is on a range of 0 to 100, with higher scores representing a better outcome.
Range of shoulder movement | 6 weeks, 3 months, 6 months, 12 months postoperatively.
  Objective measure of shoulder movement in abduction, flexion and rotation planes.
Postoperative pain score | 6 weeks
  Patient subjective pain scores following surgery. This is on a visual analogue scale, ranging from 0-10, with 10 representing more pain. Patients will be asked about their usual levels of pain on a weekly basis using the scale.
Structural integrity of repair | 6 months.
  This will be assessed by an MRI scan postoperatively to assess healing of the tear or failure of the repair.

CONTACTS AND LOCATIONS:
Overall Officials: Mrs K Rhodes, Study Director — Manchester University Foundation Trust
Locations (1):
- Manchester University Foundation NHS Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial website with more information — http://www.sstart.co.uk